CLINICAL TRIAL: NCT05827874
Title: A Randomized, Open-Label Study on the Effect of Nipocalimab on Vaccine Responses in Healthy Participants
Brief Title: A Study on the Effect of Nipocalimab on Vaccine Responses in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR109301; 2022-003131-26 (EudraCT Number); 80202135EDI1009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-04-04; First posted 2023-04-25 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Arm: (Experimental): Participants will receive Nipocalimab loading dose intravenous (IV) infusion at Week 0 followed by tetanus, diphtheria, pertussis (Tdap) and pneumococcal polysaccharide vaccine (PPSV23) vaccine challenge as an intramuscular (IM) injection on Day 3 of Week 0 and additional doses of Nipocalimab IV at Week 2 and 4.
  Interventions: Drug: Nipocalimab; Biological: Tdap; Biological: PPSV23
- Control Arm: (Other): Participants will receive PPSV23 and Tdap vaccine challenge as an IM injection on Day 3 of Week 0.
  Interventions: Biological: Tdap; Biological: PPSV23

INTERVENTIONS:
Drug: Nipocalimab — Nipocalimab will be administered as an IV infusion.
  Other Names: JNJ-80202135
  Arms: Active Arm:
Biological: Tdap — Tdap will be administered as an IM injection.
  Other Names: GSK Boostrix
Biological: PPSV23 — PPSV23 will be administered as an IM injection.
  Other Names: MSD Pneumovax23

SUMMARY:
The purpose of this study is to assess the effect of nipocalimab treatment on the antibody (a protein made in the body to response to a foreign substance) response following tetanus, diphtheria, pertussis (Tdap) vaccination in healthy participants at Week 4.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, and 12 lead electrocardiogram (ECG) performed at screening. Any abnormalities must be considered not clinically significant, and this determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening (including immunoglobulin G [IgG]). If the results of the serum chemistry panel, hematology or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participant agrees not to donate bone marrow, blood, and blood products from the study intervention administration until 3 months after receiving it
* Body mass index (BMI) between 18 and 30 kilograms per meter square (kg/m^2) (BMI = weight/height^2), inclusive, and a body weight of no less than 50 kilograms (kg)
* must be a nonsmoker (not smoked for at least 3 months prior to screening) and has not used nicotine-containing products (example, nicotine patch and vaping) for at least 3 months prior to screening
* Willing and able to adhere to the lifestyle restrictions specified in this protocol

Exclusion Criteria:

* History of liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbance
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Had major illness or surgery (example, requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from illness or surgery, or has surgery planned during the time the participant is expected to participate in the study
* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study
* Known allergies, hypersensitivity, or intolerance to pneumococcal polysaccharide vaccine (PPSV23) and tetanus, diphtheria, pertussis (Tdap) vaccines, nipocalimab, or any of their excipients
* Has a serum albumin level less than (<) 30 grams per liter (g/L) at screening or Day -1
* Has a total IgG less than or equal to (<=) 6 g/L at screening.
* Has received a tetanus (example, Tdap, Td) vaccine in the past <= 5 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with a Positive Anti-tetanus toxoid Immunoglobulin G (Anti-TT IgG) Response at 4 Weeks Post-vaccination | 4 Weeks post-vaccination at Week 0 (Up to Week 4)
  Percentage of participants with a positive anti-TT IgG response at 4 weeks post-vaccination will be reported. It is defined as pre-vaccination anti-TT IgG antibody titers are less than (<) 0.16 international units per milliliter (IU/mL) and post-vaccination anti-TT IgG titers are greater than or equal to (>=) 0.16 IU/mL, or pre-vaccination anti-TT IgG are >= 0.16 IU/mL and there is at least a 2-fold increase in post-vaccination anti-TT IgG titers.

SECONDARY OUTCOMES:
Percentage of Participants with Positive IgG Response to TT Vaccine from Baseline through 16 Weeks Post-vaccination | Baseline through 16 Weeks post-vaccination at Week 0 (Up to Week 16)
  Percentage of participants with positive IgG response to TT vaccine from baseline through 16 Weeks Post-vaccination will be reported. It is defined as pre-vaccination anti-TT IgG antibody titers are less than (<) 0.16 international units per milliliter (IU/mL) and post-vaccination anti-TT IgG titers are greater than or equal to (>=) 0.16 IU/mL, or pre-vaccination anti-TT IgG are >= 0.16 IU/mL and there is at least a 2-fold increase in post-vaccination anti-TT IgG titers.
Change from Baseline in Anti-Pneumococcal Capsular Polysaccharide (PCP) IgG Levels Over Time Through 16 Weeks Post-vaccination | Change from baseline through 16 Weeks post-vaccination at Week 0 (Up to Week 16)
  Change from baseline in anti-PCP IgG levels over time through 16 Weeks post-vaccination will be reported.
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) Through Week 16 | Up to Week 16
  Percentage of participants with TEAEs through Week 16 will be reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Percentage of Participants with Serious Adverse Events (SAEs) Through Week 16 | Up to Week 16
  Percentage of Participants with SAEs through Week 16 will be reported. A SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect, is suspected transmission of any infectious agent via a medicinal product, is medically important to prevent one of the outcomes listed above.
Percentage of Participants with Adverse Events of Special Interests (AESIs) Through Week 16 | Up to Week 16
  Percentage of participants with AESIs through Week 16 will be reported. Treatment-emergent AEs associated with the following situations are considered an AESI: a) infections that are severe or require intravenous (IV) anti-infective or operative/invasive intervention; b) hypoalbuminemia with albumin less than (<)20 grams per liter (g/L) [<] 2.0 grams per deciliter [g/dL]).
Serum Concentrations of Nipocalimab Over Time | Pre dose, 1, 24, 48, 72 hours at Week 0 and Week 2, 4, 8 and 16 post dose
  Serum concentrations of nipocalimab over time will be reported. Serum samples will be analyzed to determine concentrations of nipocalimab using a validated, specific, and sensitive immunoassay method.
Number of Participants with Anti-Drug Antibodies (ADAs) to Nipocalimab | Up to Week 16
  Number of participants with ADAs to nipocalimab will be reported.
Changes in Total IgG and its Subclasses (IgG1, IgG2, IgG3, IgG4) Serum Levels Over Time | Up to Week 16
  Changes in total IgG and its subclasses (IgG1, IgG2, IgG3, IgG4) serum levels over time will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Cossu M, Bobadilla Mendez C, Jackson A, Myshkin E, Liu G, Lam E, Beier UH, Weisel K, Scott B, Leu JH, Gao S, Dimitrova D. A randomized, open-label study on the effect of nipocalimab on vaccine responses in healthy participants. Hum Vaccin Immunother. 2025 Dec;21(1):2491269. doi: 10.1080/21645515.2025.2491269. Epub 2025 Apr 15. PMID 40232701